CLINICAL TRIAL: NCT06706115
Title: : Effect of Intranasal Breast Milk Administration on Cerebral Oxygenation, Vital Signs and Transition Time to Full Oral Feeding in Preterm Babies: Randomized Controlled Study
Brief Title: Effect of Intranasal Breast Milk Administration in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SelcukUni2545
Record Dates: First submitted 2024-05-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Newborn; Vitality; Nursing Caries; Breast Feeding
Keywords: Breast milk; Newborn Nursing; Oral Nutrition; Physiological parameters; Preterm infant
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Intervention Model Description: Randomized controlled design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal Breast Milk Group (Experimental): Preterm infants (28-37 gestation week) in the intervention group will receive 0.2 ml of breast milk intranasally three times a day for three days.
  Interventions: Other: Intranasal human breast milk
- Control Group (No Intervention): Preterm newborns in the control group will not receive any intervention.

INTERVENTIONS:
Other: Intranasal human breast milk — The information in the "Physiologic Parameter Follow-up Form" will be recorded by the investigator just 5 minutes before the intervention. The researcher will drip 0.2 ml of breast milk at room temperature (approximately 22 °C) into the nose of the infant lying in the supine position, 0.1 ml in the right nose-0.1 ml in the left nose. 5 minutes after the intervention (T1), 15 minutes after the intervention (T2) and 30 minutes after the intervention (T3), the data in the "Physiologic Parameter Follow-up Form" will be recorded by the researcher. After intranasal breast milk administration, the baby will be fed by the neonatal nurse as in routine practice. The implementation of the intervention in the study will last for three days and this process will be repeated three times every day (09.00, 12.00 and 15.00).
  Arms: Intranasal Breast Milk Group

SUMMARY:
The aim of the study was to investigate the effect of intranasal breast milk administration on cerebral oxygenation level, vital signs and time to full oral feeding in preterm infants.

DETAILED DESCRIPTION:
Breast milk is rich in pluripotent stem cells, including pluripotent stem cells that produce neuronal cells in vitro. Therefore, intranasal breast milk administration in neonates may potentially allow the transport of stem cells and other molecules into brain tissue through the nasal vasculature and permeable neonatal blood-brain barrier. In recent years, studies on intranasal breast milk administration in newborns have been published. In studies, there is evidence that intranasal breast milk may be effective in reducing cerebral damage after intracranial hemorrhage in preterm newborns and that the application can be tolerated by preterm newborns.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight >1000 gr,
* APGAR score >7 at 5 minutes after birth,
* Availability of breast milk,
* No medical diagnosis affecting cerebral oxygenation (intraventricular hemorrhage, cardiovascular and neurological disorders, anemia),
* No congenital anomalies or chromosomal abnormalities,
* No congenital anomaly (such as cleft palate) affecting nasal patency.

Exclusion Criteria:

* Being able to feed orally in all feedings
* Being fed entirely on formula milk,
* Administration of medication via the nasal route,
* Being intubated or receiving continuous positive air pressure (CPAP) support,
* Maternal substance abuse, alcohol abuse, HIV infection, untreated active tuberculosis, chemotherapy or radiotherapy treatment,
* The mother has mastitis, breast trauma, abscesses or is taking any medication that passes into the milk,
* The mother does not want to express milk.

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Infant Information Form | First measurement-First day of hospitalization
  The form developed by the researchers in line with the literature includes the identifying information of the preterm infant (gender, date of birth, gestational week at birth, mode of delivery, APGAR score, birth weight, postmenstrual age)
Physiologic Parameter Follow-up Form-Cerebral rSO2 | First measurement- 5 minutes before the intervention (T0)
  Cerebral rSO2 in the Physiological Parameter Monitoring Form will be measured 5 minutes before the intervention.
Physiologic Parameter Follow-up Form-Oxygen saturation (sPO2) | First measurement- 5 minutes before the intervention (T0)
  Oxygen saturation (sPO2) in the Physiological Parameter Monitoring Form will be measured 5 minutes before the intervention.
Physiologic Parameter Follow-up Form-Heart Rate (HR) | First measurement- 5 minutes before the intervention (T0)
  Heart rate in the Physiological Parameter Monitoring Form will be measured 5 minutes before the intervention.
Physiologic Parameter Follow-up Form-Respiratory rate | First measurement- 5 minutes before the intervention (T0)
  Respiratory rate in the Physiological Parameter Monitoring Form will be measured 5 minutes before the intervention.
Nutrition Follow-up Form-intranasal breast milk content | First measurement- intranasal breast milk content
  Intranasal breast milk content (fresh/thawed) in the Nutrition Follow-up Form will be recorded before the intervention.

SECONDARY OUTCOMES:
Physiologic Parameter Follow-up Form -Cerebral rSO2 | Second measurement- 5. minutes after the intervention (T1)
  Cerebral rSO2 in the Physiological Parameter Monitoring Form will be measured 5 minutes after the intervention.
Physiologic Parameter Follow-up Form -Cerebral rSO2 | Second measurement- 15. minutes after the intervention (T1)
  Cerebral rSO2 in the Physiological Parameter Monitoring Form will be measured 15 minutes after the intervention.
Physiologic Parameter Follow-up Form -Cerebral rSO2 | Second measurement- 30. minutes after the intervention (T1)
  Cerebral rSO2 in the Physiological Parameter Monitoring Form will be measured 30 minutes after the intervention.
Physiologic Parameter Follow-up Form -Oxygen saturation (sPO2) | Second measurement- 5. minutes after the intervention (T1)
  Oxygen saturation (sPO2) in the Physiological Parameter Monitoring Form will be measured 5 minutes after the intervention.
Physiologic Parameter Follow-up Form -Oxygen saturation (sPO2) | Second measurement- 15. minutes after the intervention (T1)
  Oxygen saturation (sPO2) in the Physiological Parameter Monitoring Form will be measured 15 minutes after the intervention.
Physiologic Parameter Follow-up Form -Oxygen saturation (sPO2) | Second measurement- 30. minutes after the intervention (T1)
  Oxygen saturation (sPO2) in the Physiological Parameter Monitoring Form will be measured 30 minutes after the intervention.
Physiologic Parameter Follow-up Form -Heart Rate (HR) | Second measurement- 5. minutes after the intervention (T1)
  Heart Rate (HR) in the Physiological Parameter Monitoring Form will be measured 5 minutes after the intervention.
Physiologic Parameter Follow-up Form -Heart Rate (HR) | Second measurement- 15. minutes after the intervention (T1)
  Heart Rate (HR) in the Physiological Parameter Monitoring Form will be measured 15 minutes after the intervention.
Physiologic Parameter Follow-up Form -Heart Rate (HR) | Second measurement- 30. minutes after the intervention (T1)
  Heart Rate (HR) in the Physiological Parameter Monitoring Form will be measured 30 minutes after the intervention.
Physiologic Parameter Follow-up Form -Respiratory rate | Second measurement- 5. minutes after the intervention (T1)
  Respiratory rate in the Physiological Parameter Monitoring Form will be measured 5 minutes after the intervention.
Physiologic Parameter Follow-up Form -Respiratory rate | Second measurement- 15. minutes after the intervention (T1)
  Respiratory rate in the Physiological Parameter Monitoring Form will be measured 15 minutes after the intervention.
Physiologic Parameter Follow-up Form -Respiratory rate | Second measurement- 30. minutes after the intervention (T1)
  Respiratory rate in the Physiological Parameter Monitoring Form will be measured 30 minutes after the intervention.
Nutrition Follow-up Form-Nutrient content | Second measurement-Nutrient content
  Nutrient content (exclusive breast milk/formula+ breast milk feeding) in the Nutrition Follow-up Form will be recorded 5 minutes after the intervention.
Nutrition Follow-up Form-Number of vomits | Second measurement- Number of vomits
  Number of vomits in the Nutrition Follow-up Form will be recorded 24 hours after the intervention.
Nutrition Follow-up Form-Number of defecations | Second measurement- Number of defecations
  Number of defecations in the Nutrition Follow-up Form will be recorded 24 hours after the intervention.
Nutrition Follow-up Form-The time of transition to full oral feeding | Second measurement- The time of transition to full oral feeding
  The time of transition to full oral feeding, which is found on the Feeding Follow-up Form, will be monitored and recorded in medical records until the baby is discharged.
Nutrition Follow-up Form-Discharge time | Second measurement- Discharge time
  Discharge time, which is found on the Feeding Follow-up Form, will be monitored and recorded in medical records until the baby is discharged.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kucukoglu, Prof, Principal Investigator — Selcuk University
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Keller T, Korber F, Oberthuer A, Schafmeyer L, Mehler K, Kuhr K, Kribs A. Intranasal breast milk for premature infants with severe intraventricular hemorrhage-an observation. Eur J Pediatr. 2019 Feb;178(2):199-206. doi: 10.1007/s00431-018-3279-7. Epub 2018 Nov 1. PMID 30386923
- [Background] Hoban R, Gallipoli A, Signorile M, Mander P, Gauthier-Fisher A, Librach C, Wilson D, Unger S. Feasibility of intranasal human milk as stem cell therapy in preterm infants with intraventricular hemorrhage. J Perinatol. 2024 Nov;44(11):1652-1657. doi: 10.1038/s41372-024-01982-8. Epub 2024 Apr 30. PMID 38688998
- [Background] Muelbert M, Alexander T, Pook C, Jiang Y, Harding JE, Bloomfield FH. Cortical Oxygenation Changes during Gastric Tube Feeding in Moderate- and Late-Preterm Babies: A NIRS Study. Nutrients. 2021 Jan 25;13(2):350. doi: 10.3390/nu13020350. PMID 33503882
- [Background] Yucel A, Kucukoglu S, Soylu H. The Effect of Breast Milk Odor on Feeding Cues, Transition Time to Oral Feeding, and Abdominal Perfusion in Premature Newborns: A Randomised Controlled Trial. Biol Res Nurs. 2024 Jan;26(1):160-175. doi: 10.1177/10998004231200784. Epub 2023 Sep 8. PMID 37682253
- [Derived] Yucel A, Kucukoglu S, Konak M. The Effect of Intranasal Breast Milk Administration on Cerebral Oxygenation, Vital Signs and Time to Full Oral Feeding in Preterm Infants: a Randomised Controlled Study Protocol. Nurs Crit Care. 2026 Jan;31(1):e70262. doi: 10.1111/nicc.70262. PMID 41542903